CLINICAL TRIAL: NCT02747355
Title: Expression of Different Proliferation Biomarkers in Adreno-cortical Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, leonard.saiegh, M.D., Bnai Zion Medical Center
Other Study IDs: BnaiZion
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Adrenal Cortex Neoplasms; Adrenal Cortex Diseases
MeSH Terms: conditions — Adrenal Cortex Neoplasms; Adrenal Cortex Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — adrenal tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
In adrenal tumors, the investigators will examine if there is any correlation between WIESS criteria, prognosis of the tumor, and the different labeling index of the following proliferation biomarkers: MCM3, MCM2, KI-67, P53, NEUROPILIN -1, METALLOTHIONEIN, SEMAPHORIN-3A.

DETAILED DESCRIPTION:
One of the problems in managing adrenocortical tumors is the ability to distinguish between benign and malignant tumors, while needle biopsy is unable to distinguish between the two situations. Therefore, when imaging tests demonstrate a suspected malignant adrenal tumor, surgical excision of the tumor is needed. Usually, the histological WIESS criteria are used in order to determine malignancy. However, there are cases when adrenal tumors were defined by WIESS criteria as benign but metastasized later. Moreover, there is no reliable test than can determine prognosis. KI-67 labeling index is a proliferation biomarker which is used to tell more about the malignant potential and prognosis of adrenal carcinoma.

In various types of tumors, proliferation biomarkers are used in attempt to tell about prognosis. In this study, the investigators will examine whether some biomarkers can differentiate between adrenal carcinoma and adenoma and if the degree of expression of these markers is correlated with prognosis.

The investigators will retrospectively collect 30 cases of adrenal carcinoma, 30 cases of adrenal adenoma and 10 cases of normal adrenals. All specimens are preserved with formalin. The investigators will re-review the WIESS criteria and all samples will be analyzed for the index labeling of the following proliferation biomarkers: MCM3, MCM2, KI-67, P53, NEUROPILIN -1, METALLOTHIONEIN, SEMAPHORIN-3A. The investigators will examine if there is any correlation between the labeling index of each biomarker, WIESS criteria and prognosis of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* adrenal carcinoma
* adrenal adenoma
* normal adrenal tissue

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adrenal tissue from patients diagnosed with adrenocortical carcinoma, adrenal adenoma and normal adrenals from patients who had renal and adrenal excision for renal cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-08-18 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
MCM3 expression | 1 year
  Difference in MCM3 labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
MCM2 expression | 1 year
  Difference in MCM2 labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
P53 expression | 1 year
  Difference in P53 labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
NEUROPILIN -1 expression | 1 year
  Difference in NEUROPILIN -1 labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
METALLOTHIONEIN expression | 1 year
  Difference in METALLOTHIONEIN labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
SEMAPHORIN-3A expression | 1 year
  Difference in SEMAPHORIN-3A labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
E-caderein expression | 1 year
  Difference in E-caderein labeling index between adrenal cortical adenoma versus adrenocortical carcinoma

SECONDARY OUTCOMES:
KI67 | 1 year
  Difference in Ki67 labeling index between adrenal cortical adenoma versus adrenocortical carcinoma
Prognosis | 1 year
  Correlation between the labeling index of each biomarker, WIESS criteria and prognosis of the tumor.

IPD SHARING:
Plan to Share IPD: Yes